CLINICAL TRIAL: NCT05493007
Title: The Efficacy and Safety of Sandbag Self Walking-MSAT on Inpatients With Acute Low Back Pain Caused by Traffic Accidents: A Randomized Controlled Trials
Brief Title: The Efficacy and Safety of Sandbag Self Walking-MSAT on Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-10
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sandbag motion style acupuncture treatment (Experimental): The MSAT group will recieve 3 sessions of MSAT; on second, third, fourth day after hospitalization.
  A trained doctor of Korean medicine with at least 3 years of clinical experience will conduct the MSAT.
  The MSAT group will be also treated with other Korean medical treatment everyday: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Sandbag motion style acupuncture treatment; Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group will be received Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine
  Interventions: Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Sandbag motion style acupuncture treatment — Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation.
  Arms: Sandbag motion style acupuncture treatment
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine.

SUMMARY:
This study is a double blind, randomized controlled trail. condition/disease: acute low back pain treatment/intervention: motion style acupuncture treatment

DETAILED DESCRIPTION:
Motion Style Acupuncture Treatment(MSAT) is a therapeutic technique using acupuncture needle created in Jaseng Hospital. This treatment involves patients with musculoskeletal pain to move the part of their body actively during acupuncture treatment under physicians' observation. This treatment is known to relieve the pain and increase the range of motion(ROM). However, there has been no specific value for the effect of this treatment.

So, the investigators conducted a randomized controlled trials to verify the efficacy and safety of Sandbag MSAT. From June 2021 to June 2023, the investigators collected 104 inpatients who were suffered from Low back pain with the numeric rating scale(NRS) over 5 after injury by acute traffic accident(TA). For experimental group(n=52), the investigators conducted MSAT three times(on 2nd, 3rd and 4th day of hospitalization) and other Korean medical treatment. For control group(n=52), just Korean medical treatment except MSAT was conducted. For these two groups, the investigators compared NRS, Visual Analogue Scale(VAS), Range Of Motion(ROM), the amount of pain via NRS(Numeric Rating Scale), VAS(Visual Analogue Scale), ROM(Range Of Motion), Oswestry Disability Index (ODI), and EuroQol 5-Dimension (EQ-5D), EuroQol Visual Analogue Scale (EQ-VAS), Short Form-12 Health Survey version 2, SF-12 v2), The Posttraumatic Stress Disorder Checklist for DSM-5(PCL-5-K), Patient Global Impression of Change (PGIC).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years on the date they sign the consent form
* Patients who needs hospitalization due to acute low back pain that occurred within 7 days after traffic accident
* Patients with NRS ≥ 5 for low back pain
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients with a specific serious disease that may cause spinal pain: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms
* Patients who have had surgery or procedures within the last three weeks
* The cause of pain is due to soft tissue disease, not the spine: tumors, fibromyalgia, rheumatoid arthritis, gout, etc.
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* If acupuncture is inadequate or unsafe: patients with hemorrhagic, receiving anticoagulants, severe diabetes and cardiovascular disease
* Patients who are pregnant or planning to become pregnant
* Patients with a serious mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of Low back pain | Change from baseline NRS at 4 days
  The extent of Low back pain and discomfort will be assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their low back pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of Low back pain | visit2(day2), visit3(day3), visit4(day4), day of discharge(up to 14days)
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Numeric Rating Scale(NRS) of leg pain | visit1(day1), visit2(day2), visit3(day3), visit4(day4), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their leg pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual Analogue Scale (VAS) of leg pain | visit2(day2), visit3(day3), visit4(day4), day of discharge(up to 14days)
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Physical examination (Lumbar range of motion) | visit2(day2), visit3(day3), visit4(day4), day of discharge(up to 14days)
  ROM of flexion, extension, lateral flexion, rotation will be measured.
Oswestry Disability Index (ODI) | visit2(day2), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  The Oswestry Disability Index (ODI) is a 10-item questionnaire that measures a patient's self-reported Low back pain related disability.
EuroQol 5-Dimension (EQ-5D) | visit2(day2), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
EuroQol Visual Analogue Scale (EQ-VAS) | visit2(day2), day of discharge(up to 14days)
  he EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Short Form-12 Health Survey version 2 (SF-12 v2) | visit2(day2), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  SF-12v2 Health Survey is a practical, reliable, and valid measure of physical and mental health. It assesses the same eight health domains as the SF-36v2 with one or two questions per domain: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health.
Patient Global Impression of Change (PGIC) | visit2(day2), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5-K) | visit2(day2), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD, making a provisional PTSD diagnosis.
Adverse events | visit2(day2), visit3(day3), visit4(day4), day of discharge(up to 14days), visit6(1 month after discharge), visit7(3 months after discharge)
  Check adverse events every visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No